CLINICAL TRIAL: NCT00000273
Title: A Laboratory Model for Heroin Abuse Medications
Brief Title: A Laboratory Model for Heroin Abuse Medications - 8
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #4857/5982R; 5P50DA009236-18 (NIH)
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Heroin Dependence; Opioid-Related Disorders; Substance-Related Disorders
Keywords: heroin, opioid disorders, substance related disorders
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders; Substance-Related Disorders | interventions — Opiate Alkaloids; Morphine; Fentanyl; Buprenorphine; Oxycodone; Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Opiates (Experimental): Opiate-dependent individuals who were currently not seeking treatment for their drug use, completed the 6-week protocol.
  Interventions: Drug: opiates

INTERVENTIONS:
Drug: opiates — prescription opioids
  Other Names: morphine; fentanyl; buprenorphine; oxycodone; methadone

SUMMARY:
The purpose of this study is to evaluate the effects of treatment medications (methadone, buprenorphine, LAAM, naltrexone, naltrexone microcapsules, and methoclocinnamox) on I.V. and smoked heroin self-administration."

DETAILED DESCRIPTION:
Abuse of prescription opioid medications has increased dramatically in the U.S. during the past decade, as indicated by a variety of epidemiological sources. However, few studies have systematically examined the relative reinforcing effects of commonly abused opioid medications. The current inpatient study was designed to compare the effects of intravenously delivered fentanyl , oxycodone, morphine, buprenorphine and heroin in morphine-maintained heroin abusers. All of the participants received all of the drugs tested; drugs and doses were administered in non-systematic order.

ELIGIBILITY:
Inclusion Criterion

1. DSM IV criteria for opioid dependence
2. No major mood, psychotic, or anxiety disorder
3. Physically healthy
4. Able to perform study procedures
5. 21-45 years of age
6. Current use of i.v. heroin in amounts/frequencies
7. Not seeking treatment for opioid dependence

Exclusion Criterion

1. DSM IV criteria for dependence on drugs other
2. Participants requesting treatment
3. Participants on parole or probation
4. Pregnancy or lactation
5. Birth, miscarriage or abortion with 6 months
6. Recent history of or current significant violent behavior
7. Current major Axis I psychopathology, other than heroin dependence ( e.g., mood disorder with functional impairment or suicide risk, schizophrenia), which might interfere with ability to participate in the study
8. Hepatitis with SGOT or SGPT > 3 times normal
9. Significant suicide risk
10. Current or history of chronic pain
11. Sensitivity, allergy, or contraindication to opioids

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 1995-08; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Amount drug self-administered | 90 minutes
  All of the participants received all of the drugs tested; drugs and doses were administered in non-systematic order. Participants were instructed to choose between the dose that they had received during the sample session or another reward..

SECONDARY OUTCOMES:
Subjective responses | 90 min
  Four questionnaires were used to assess subjective effects

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Kleber, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - New York State Psychiatric Institute, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Comer SD, Sullivan MA, Whittington RA, Vosburg SK, Kowalczyk WJ. Abuse liability of prescription opioids compared to heroin in morphine-maintained heroin abusers. Neuropsychopharmacology. 2008 Apr;33(5):1179-91. doi: 10.1038/sj.npp.1301479. Epub 2007 Jun 20. PMID 17581533